CLINICAL TRIAL: NCT03300310
Title: Impact of the Nurse Visit on Observance of the Intake of Oral Carcinological Treatment
Brief Title: Impact of the Nurse Visit on Observance of the Intake of Oral Carcinological Treatment in the Elderly
Acronym: IPIO-PA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Despite an extension of the planned duration of inclusion and an enrolled patient number inferior than planned, coordinating investigator considered that it was more reasonable to stop inclusions in order to analyze the data already available
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC17_0096; 2017-A00629-44 (Registry Identifier: ANSM)
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Oncology, Gerontology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with nursing visit (Experimental): a nurse visit is scheduled twice a week during 3 months at patient home.
  Interventions: Other: nursing visit
- without nursing visit (Experimental): no nursing visit
  Interventions: Other: no nursing visit

INTERVENTIONS:
Other: nursing visit — nursing visit at patient home
  Arms: with nursing visit
Other: no nursing visit — the patient take his treatment without nursing visit
  Arms: without nursing visit

SUMMARY:
The increasingly used oral anticancer treatments allow the patient to reduce treatment and social constraints to reduce hospitalization costs. The counterpart is a decrease in the monitoring of the correct intake of drugs and the detection of side effects. These two risks are major in the elderly, due to comorbidities, poly-medication and decreased attention. The project objective to evaluate the impact of a bi-weekly nursing visit to the patients' homes for 3 months, compared to a conventional management without a nursing visit. It is a prospective, randomized, controlled, multicenter study to include 224 patients over 18 months. The impact will be assessed by counting the tablets not taken and by filling an observation booklet with the nurse at home.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 70 and over
* Patient initiating an oral anticancer treatment (Chemotherapy, Targeted therapy, 2nd generation hormone therapy type Acetate abiraterone and Enzalutamide)
* Patient who received an onco-geriatric assessment
* Patient with informed consent signed

Exclusion Criteria:

* Patient in a medical institution
* Patient under exclusive hormone therapy
* Patient already eligible for nurse support
* Patient not speaking French
* Patient under tutelage and guardianship or under safeguard of justice
* Patient already included in a research protocol
* Patient sharing his or her home with a person receiving nursing care at home more than once a week and for a period longer than 1 month after the patient's inclusion.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Comparison, at 3 months after the oncological treatments began, of the observance rate of the anticancer drugs (corresponding to the entire carcinological protocol) with or without passage of a nurse at the patient's home. | 3 months

SECONDARY OUTCOMES:
Comparison of the patient's perception of observance to anticancer therapy | 3 months
Comparison of causes of possible premature and definitive cessation of cancer treatments 3 months after the start of treatment and changes in treatment (dose, rhythm of cycles) | 3 months
Assessment of patients' satisfaction (of the arm with passage of the nurse) and the professionals | 3 months
Determination of the percentage of patients able to be included in the study compared to the number of patients who received an oncogeriatric assessment | 3 months

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - ICO Angers, Angers
  - CHD Vendée, La Roche-sur-Yon
  - CHU de Nantes, Nantes
  - Hôpital privé du Confluent, Nantes
  - ICO Nantes, Saint-Herblain
  - CH Saint Nazaire, Saint-Nazaire

IPD SHARING:
Plan to Share IPD: No